CLINICAL TRIAL: NCT01131130
Title: A Study to Evaluate the Product Feasibility of a New Silicone Hydrogel Lens
Brief Title: Feasibility of a New Silicone Hydrogel Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 655
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-03

CONDITIONS: Myopia
Keywords: Contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Investigational contact lens (Experimental): Bausch & Lomb
  Interventions: Device: Investigational contact lens
- Acuvue Oasys Contact Lens (Active Comparator): Johnson & Johnson Lens
  Interventions: Device: Acuvue Oasys Contact Lens
- Air Optix Aqua (Active Comparator): Ciba Vision
  Interventions: Device: Air Optix Aqua

INTERVENTIONS:
Device: Investigational contact lens — After one week of wearing the first lens type, the participants will crossover to the second lens type for one week, and then crossover to the third lens type.
  Arms: Investigational contact lens
Device: Acuvue Oasys Contact Lens — After one week of wearing the first lens type, the participants will crossover to the second lens type for one week, and then crossover to the third lens type.
  Arms: Acuvue Oasys Contact Lens
Device: Air Optix Aqua — After one week of wearing the first lens type, the participants will crossover to the second lens type for one week, and then crossover to the third lens type.
  Arms: Air Optix Aqua

SUMMARY:
The objective of this study is to determine the product feasibility of the investigational contact lens (Test) when compared to the currently marketed Acuvue Oasys contact lens (Control) and the Air Optix Aqua contact lens (Control) when worn by adapted wearers of soft contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have clear central corneas and be free of any anterior segment disorders.
* Participants must be adapted wearers of soft contact lenses, wear a lens in each eye, and each lens must be of the same manufacture and brand.
* Participants must be myopic and require lens correction from -0.75 D to - 4.75D in each eye.

Exclusion Criteria:

* Participants who have worn gas permeable (GP) contact lenses within the last 30 days or who have worn polymethylmethacrylate (PMMA) lenses within the last three months.
* Participants with any systemic disease affecting ocular health.
* Participants using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Participants with an active ocular disease or are using any ocular medication.
* Participants who have had any corneal surgery (eg, refractive surgery).
* Participants who are allergic to any component in the study care products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Carains, MCOptom, PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 120 participants enrolled in this bilateral eye, three-period crossover study at four investigative sites in the United States (US). All participants were adapted wearers of soft contact lenses. The first participant was enrolled in the study on 5/10/2010 and the last participant exited the study on 6/10/2010.
Pre-assignment Details: Participants were equally randomized to one of six treatment sequences of the investigational RD2106 contact lens (Test), the Air Optix Aqua contact lens, and the Acuvue Oasys contact lens. Of the 120 participants enrolled 2 were ineligible at baseline and 2 discontinued following dispensing of lenses. 116 participants completed the study.
Groups:
- Over All Study: Participants were equally randomized to one of six treatment sequences of the investigational RD2106 contact lens (Test), the Air Optix Aqua contact lens, and the Acuvue Oasys contact lens. Crossover occurred following 1 week of lens wear. The 6 groups were as follows Test, Air Optix Aqua, Acuvue Oasys; Test, Acuvue Oasys, Air Optix Aqua; Air Optix Aqua, Test, Acuvue Oasys; Air Optix Aqua, Acuvue Oasys, Test; Acuvue Oasys, Test, Air Optix Aqua; Acuvue Oasys, Air Optix Aqua, Test.
Period: Period 1 - Baseline
Arm/Group | Over All Study
Started | 118
Completed | 117 (Participant was discontinued 1 day following dispensing and not reported in result tables)
Not Completed | 1
Not completed — Pregnancy | 1
Period: Period 2 - Crossover
Arm/Group | Over All Study
Started | 117
Completed | 117
Not Completed | 0
Period: Period 3- Crossover
Arm/Group | Over All Study
Started | 117
Completed | 116
Not Completed | 1
Not completed — + Slit lamp finding | 1

BASELINE CHARACTERISTICS:
Population: All eligible, dispensed participants
Arm/Group | Over All Study
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 117

OUTCOME MEASURES:

1. Secondary Outcome: Lens Wettability, Test Lens vs. Acuvue Oasys
Description: Lens wettability was assessed at each visit as Grade 4 - 0, with 4=optimal (100% of anterior surface wettable) and 0=severe (Presence of one or more non-wetting areas > 0.5 mm in size).
Time Frame: 7 days
Population: All eligible, dispensed eyes
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Contact Lens | Acuvue Oasys Contact Lens
Number analyzed (Participants) | 115 | 116
Number analyzed (eyes) | 229 | 232
eyes
  Optimal | 210 | 214
  Slight | 14 | 16
  Mild | 1 | 0
  Moderate | 3 | 2
  Severe | 1 | 0

2. Primary Outcome: Comfort Throughout the Day - Test Lens vs. Air Optix Aqua Lens
Description: Subjective measurements of lens comfort were rated on a scale from 0 to 100, where 100 was the most favorable.
Time Frame: 7 days
Population: All eligible dispensed eyes
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Investigational Contact Lens | Air Optix Aqua
Number analyzed (Participants) | 115 | 116
Number analyzed (eyes) | 230 | 232
units on a scale | 74.3 (22.1) | 79.4 (22.1)

3. Primary Outcome: Comfort Throughout the Day - Test Lens vs. Acuvue Oasys
Description: Subjective measurements of lens comfort were rated on a scale from 0 to 100, where 100 was the most favorable.
Time Frame: 7 days
Population: All eligible, dispensed eyes
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Investigational Contact Lens | Acuvue Oasys Contact Lens
Number analyzed (Participants) | 115 | 116
Number analyzed (eyes) | 230 | 232
units on a scale | 74.3 (22.1) | 88.0 (22.1)

4. Secondary Outcome: Lens Wettability, Test Lens vs. Air Optix Aqua
Description: as for outcome 1
Time Frame: 7 days
Population: All eligible, dispensed eyes
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Contact Lens | Air Optix Aqua
Number analyzed (Participants) | 115 | 116
Number analyzed (eyes) | 229 | 231
eyes
  Optimal | 210 | 219
  Slight | 14 | 10
  Mild | 1 | 0
  Moderate | 3 | 2
  Severe | 1 | 0

ADVERSE EVENTS:
Time Frame: 7 Days
Arm/Group | Investigational Contact Lens | Acuvue Oasys Contact Lens | Air Optix Aqua
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/117 | 0/117
Other Adverse Events (participants affected / at risk) | 0/117 | 0/117 | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other